CLINICAL TRIAL: NCT00643539
Title: Multicenter, Open, Randomized Comparative Trial To Compare Bacteriological And Clinical Efficacy Of Azithromycin Versus Amoxicillin In Children With Streptococcus Tonsillitis
Brief Title: Multicenter, Open, Randomized Comparative Trial To Compare The Efficacy Of Azithromycin Versus Amoxicillin In Children With Strep Throat
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0661037
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Tonsillitis
MeSH Terms: conditions — Tonsillitis | interventions — Azithromycin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Clamoxyl
- 2 (Experimental)
  Interventions: Drug: Zithromax

INTERVENTIONS:
Drug: Zithromax — azithromycin (Zithromax) pediatric suspension formulation (200 mg/5 ml) administered as an oral suspension at a dose of 20 mg/kg once a day (maximal dose 500 mg/day) for 3 consecutive days
  Arms: 2
Drug: Clamoxyl — Amoxicillin (Clamoxyl) pediatric formulation (500 mg/5 ml) administered as an oral suspension at a dose of 25 mg/kg twice daily (maximal dose 2 g/day) for 6 consecutive days
  Arms: 1

SUMMARY:
The primary objective was to compare the bacteriological efficacy at Day 10 of azithromycin pediatric suspension (20 mg/kg/day once daily for 3 consecutive days) versus amoxicillin pediatric suspension (50 mg/kg/day in 2 doses for 6 consecutive days) in children aged 3-15 years with Group A streptococcal acute pharyngitis/tonsillitis. Secondary objectives were assessments of bacteriological efficacy at Day 30 and clinical efficacy at Day 10 and Day 30.

ELIGIBILITY:
Inclusion Criteria:

Outpatients with an acute pharyngitis erythematous or erythematopultaceous with modification of pharynx aspect and fever of ≥38° C, and patients either with or without spontaneous pharyngeal pain or upon swallowing and enlargement of the cervical lymph node (mandibular area) were eligible for inclusion. All subjects should have had a positive rapid strep test and a positive culture for Group A beta-hemolytic streptococcus.

Exclusion Criteria:

Patients with pseudomembranous, vesicular, ulcerous or ulceronecrotic pharyngitis were excluded.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2002-12; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Bacteriologic success (Eradication: elimination of the original GABS; or Colonization: elimination of the original GABS but isolation of another stain of GABS) or failure (Persistence: presence of original GABS on repeated culture samples) rate | Day 10

SECONDARY OUTCOMES:
Bacteriological success or failure rate | Day 30
Clinical success (resolution of signs and symptoms, or sufficient improvement; no additional antibacterial therapy indicated) or failure (insufficient improvement or worsening of signs and symptoms; additional antibacterial therapy indicated) rate | Day 10
Clinical success or failure rate | Day 30
Serious and non-serious adverse events (AEs) rates | continuous
Rate of poststreptococcal complications and new disease occurrence since Day 10 | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- France (38):
  - Pfizer Investigational Site, Ancenis
  - Pfizer Investigational Site, Asnières-sur-Seine
  - Pfizer Investigational Site, Auch
  - Pfizer Investigational Site, Boulogne
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Brivé
  - Pfizer Investigational Site, Cannes LA BOCA
  - Pfizer Investigational Site, Chambéry
  - Pfizer Investigational Site, Champigny-sur-Marne
  - Pfizer Investigational Site, Châlons-en-Champagne
  - Pfizer Investigational Site, Combs-la-Ville
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Draguignan
  - Pfizer Investigational Site, Essey-lès-Nancy
  - Pfizer Investigational Site, Lagny
  - Pfizer Investigational Site, Les Sables-d'Olonne
  - Pfizer Investigational Site, Les Ulis
  - Pfizer Investigational Site, Levallois-Perret
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Massy
  - Pfizer Investigational Site, Meudon-la-Forêt
  - Pfizer Investigational Site, Meysieu
  - Pfizer Investigational Site, Millery
  - Pfizer Investigational Site, Nogent-sur-Marne
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Saint-Marcel
  - Pfizer Investigational Site, Saint-Quentin
  - Pfizer Investigational Site, Salon-de-Provence
  - Pfizer Investigational Site, Sartrouville
  - Pfizer Investigational Site, Sélestat
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Thionville
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Tresses
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
  - Pfizer Investigational Site, Varois-et-Chaignot
  - Pfizer Investigational Site, Vence
  - Pfizer Investigational Site, Versailles

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661037&StudyName=Multicenter%2C%20Open%2C%20Randomized%20Comparative%20Trial%20To%20Compare%20The%20Efficacy%20Of%20Azithromycin%20Versus%20Amoxicillin%20In%20Children%20With%20Strep%20Throat